CLINICAL TRIAL: NCT06265012
Title: A Phase 1 Randomized, Single-Blind, Placebo-Controlled, Ascending Dose Study to Evaluate the Safety and Immunogenicity of rVSV∆G-MARV-GP [Angola] (PHV01, MARV GP Vaccine) in Healthy Adults
Brief Title: Study to Evaluate the Recombinant VSV (rVSV)-Marburg Virus Vaccine Candidate (PHV01) in Healthy Adult Subjects
Acronym: PHV01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Public Health Vaccines LLC (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PHV01-C-101
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Marburg Virus Disease
Keywords: live, attenuated vaccine; Marburg virus; PHV01 (rVSV-MARV GP) vaccine; recombinant vesicular stomatitis virus
MeSH Terms: conditions — Marburg Virus Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A, Low Dose PHV01 (Experimental): Group A (10 subjects) PHV01 @ 10^5 pfu/dose given once
  Interventions: Biological: PHV01
- Group B, Medium Dose PHV01 (Experimental): Group B (10 subjects) PHV01 @ 10^6 pfu/dose given once
  Interventions: Biological: PHV01
- Group C, Hjigh Dose PHV01 (Experimental): Group C (10 subjects) PHV01 @ 10^7 pfu/dose given once
  Interventions: Biological: PHV01
- Group D, Placebo (Placebo Comparator): Group D (6 subjects) Placebo given once
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PHV01 — Marburg virus vaccine
  Arms: Group A, Low Dose PHV01; Group B, Medium Dose PHV01; Group C, Hjigh Dose PHV01
Biological: Placebo — Lactated Ringer's Solution
  Arms: Group D, Placebo

SUMMARY:
This is a Phase 1 randomized, single-blind, placebo-controlled, ascending dose study to evaluate the safety and immunogenicity of rVSV∆G-MARV-GP [Angola] (PHV01, Marburg Virus glycoprotein [MARV GP] Vaccine) in healthy adults. PHV01 is a live, attenuated rVSV vaccine expressing the MARV GP. The main questions it aims to answer are:

* Which dose of PHV01 is safe to administer to, and well-tolerated by healthy adult subjects?
* What is the immunologic response (Marburg-specific Immunoglobulin G (IgG) ELISA antibody and neutralizing antibodies) to each dose level?

Participants will receive 1 intramuscular injection of PHV01 or placebo on Day 1 and will be followed for 181 days.

DETAILED DESCRIPTION:
Participants will be randomly assigned to vaccine or placebo in four dose cohorts, starting with evaluation of safety using a sentinel group at each dose level, followed by dosing of the rest of the group in the next cohort. That next cohort will also dose the sentinel group with the next higher dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or non-pregnant, non-lactating females, age 18-60 years
* Given written informed consent
* No clinically significant health problems
* Negative test for SARS-CoV-2
* Agree to avoid conception through Day 29
* Agree to minimize blood and body fluid exposures to others after vaccination through Day 29
* Agree to avoid exposure to immunocompromised persons after vaccination through Day 29

Exclusion Criteria:

* Prior infection with Marburg virus, related filovirus, or Ebola virus
* Prior infection with vesicular stomatitis virus (VSV)
* Received any VSV-vectored vaccine
* BMI of ≥ 35
* Household contact who is immunodeficient, or on immunosuppressive medication
* Hepatitis B, hepatitis C, HIV-1, HIV-2, history of long COVID, diabetes, atopic dermatitis (eczema), chronic inflammatory disease, autoimmune or autoinflammatory disorder, malignancy, chronic or active neurologic disorder
* History of severe reactions to any vaccine or history of severe allergies
* Receipt of investigational product up to 30 days prior to randomization
* Receipt of licensed or authorized non-live vaccines within 14 days of planned study immunization (30 days for live vaccines).
* Known allergy to components of PHV01
* Injection sites obscured by tattoos or physical condition
* Significant psychiatric or medical condition or laboratory abnormality on screening
* History of Guillain Barre Syndrome or any chronic or acute neurological disorder
* Alcohol or illicit drug abuse within past 5 years
* Pregnant or lactating female
* Administration of blood or IgG within 60 days preceding study
* Administration of systemic chronic immunosuppressants (defined as more than 14 days) or other immune modifying drugs within 6 months of study entry
* History of blood donation within 60 days of study
* Unwilling to undergo diagnostic evaluation of rash (skin biopsy, if indicated) or joint symptoms (arthrocentesis if indicated by joint effusion), in both cases if acceptable to subject
* Elective surgery planned during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Solicited Adverse Events (AEs) | Study Days 1-15
  Incidence and severity of solicited injection site [(arm pain, local tenderness, erythema (redness), and induration (swelling/firmness)] and systemic AEs
Unsolicited AEs | Study Days 1-29
  Incidence and severity of unsolicited AEs
Other AEs | Study Days 1-181
  Incidence and severity of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) and Medically Attended Adverse Events (MAAEs)
Immunogenicity, Antibodies (Ab) | Injection through 28 days
  Geometric mean titers (GMT) of Marburg GP protein-specific IgG antibody as measured by enzyme-linked immunosorbent assay (ELISA) on days 1 and 29
Immunogenicity, Neutralizing antibodies (NEUT) | Injection through 28 days
  PsVNT50 and PsVNT80 MARV GP-specific neutralizing antibodies titers

CONTACTS AND LOCATIONS:
Overall Officials: Joan Fusco, PhD, Study Chair — Public Health Vaccines; Richard Kenney, MD, Study Director — Public Health Vaccines
Locations (1):
- CenExel RCA, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT06265012/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT06265012/SAP_001.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT06265012/ICF_002.pdf